CLINICAL TRIAL: NCT00953134
Title: Periconceptional Iron Supplementation on Iron and Folate Indicators Among Pregnant and Non-pregnant Women in Rural Bangladesh.
Brief Title: Periconceptional Iron Supplementation in Rural Bangladesh
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Periconceptional_Fe
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: periconceptional; iron; folic acid; supplementation
MeSH Terms: conditions — Anemia | interventions — ferrous fumarate; Iron; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IFA - Iron and Folic Acid (60 mg of ferrous fumarate and 400 mcg folic acid)
  Interventions: Dietary Supplement: Ferrous fumarate (iron); Dietary Supplement: folic acid
- 2 (Active Comparator): FA - Folic Acid (400 mcg folic acid)
  Interventions: Dietary Supplement: folic acid

INTERVENTIONS:
Dietary Supplement: Ferrous fumarate (iron) — 60 mg of ferrous fumarate
  Other Names: Powdered micronutrient supplement (Sprinkles®, Ped-Med Ltd)
  Arms: 1
Dietary Supplement: folic acid — 400 mcg folic acid
  Other Names: Powdered micronutrient supplement (Sprinkles®, Ped-Med Ltd)

SUMMARY:
The investigators hypothesize that periconceptional iron supplementation to married, nulliparous women in rural Bangladesh will significantly reduce anemia and improve hemoglobin concentrations before and during pregnancy.

DETAILED DESCRIPTION:
In 2007, the National Strategy for Anemia Prevention and Control in Bangladesh included adolescents and newly married women as target groups for future iron and folic acid (IFA) supplementation programs. This double-blinded RCT examined the effect of daily periconceptional IFA vs. folic acid (FA) on anemia and iron indictors before and during pregnancy among married, nulliparous women in rural Bangladesh. Biochemical indices were collected at baseline and either at 15 weeks gestation or after 9 months among non-pregnant women (NPW).

ELIGIBILITY:
Inclusion Criteria:

Women were eligible if they were:

* Married
* Nulliparous
* < 40 years old
* Living in the same household as their husband

Exclusion Criteria:

Women were excluded if they were:

* Pregnant at enrollment
* Planning to move out of the region
* Using iron supplements within the previous 3 months
* Using an implant form of birth control, or had surgery to prevent pregnancy
* Women with a Hb concentration of < 70 g/L, defined as severely anemic according to WHO definition (5), were excluded from the study and appropriately treated

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 273 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | February 2007-February 2008

SECONDARY OUTCOMES:
Plasma ferritin | February 2007-February 2008

CONTACTS AND LOCATIONS:
Overall Officials: Amina Khambalia, MSc, Study Director — The Hospital for Sick Children
Locations (1):
- Brac, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Derived] Khambalia AZ, O'Connor DL, Macarthur C, Dupuis A, Zlotkin SH. Periconceptional iron supplementation does not reduce anemia or improve iron status among pregnant women in rural Bangladesh. Am J Clin Nutr. 2009 Nov;90(5):1295-302. doi: 10.3945/ajcn.2009.28350. Epub 2009 Sep 30. PMID 19793860